CLINICAL TRIAL: NCT01157364
Title: An Open-label (Stage 1) and Randomized (Stage 2), 24 Month Study of Safety and Efficacy of Bimatoprost Drug Delivery System in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Efficacy of a New Ophthalmic Formulation of Bimatoprost in Patients With Open Angle Glaucoma and Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-041D; 2011-005091-42 (EudraCT Number)
Record Dates: First submitted 2010-07-02; First posted 2010-07-07 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- bimatoprost 20 µg generation 2, bimatoprost 0.03% (Other): Single dose of bimatoprost ophthalmic 20 µg generation 2 administered in the study eye on Day 1. One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
  Interventions: Drug: bimatoprost 20 µg generation 2; Drug: bimatoprost 0.03%
- bimatoprost 15 µg generation 2, bimatoprost 0.03% (Other): Single dose of bimatoprost ophthalmic 15 µg generation 2 administered in the study eye on Day 1, and once between 90 days and 12 months after the first dose (if applicable). One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
  Interventions: Drug: bimatoprost 15 µg generation 2; Drug: bimatoprost 0.03%
- bimatoprost 10 µg generation 2, bimatoprost 0.03% (Other): Single dose of bimatoprost ophthalmic 10 µg generation 2 administered in the study eye on Day 1, and once between 90 days and 12 months after the first dose (if applicable). One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
  Interventions: Drug: bimatoprost 10 µg generation 2; Drug: bimatoprost 0.03%
- bimatoprost 6 µg generation 2, bimatoprost 0.03% (Other): Single dose of bimatoprost ophthalmic 6 µg generation 2 administered in the study eye on Day 1, and once between 90 days and 12 months after the first dose (if applicable). One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
  Interventions: Drug: bimatoprost 6 µg generation 2; Drug: bimatoprost 0.03%
- bimatoprost 15 µg generation 1, bimatoprost 0.03% (Other): Single dose of bimatoprost ophthalmic 15 µg generation 1 administered in the study eye on Day 1. One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
  Interventions: Drug: bimatoprost 15 µg generation 1; Drug: bimatoprost 0.03%
- bimatoprost 10 µg generation 1, bimatoprost 0.03% (Other): Single dose of bimatoprost ophthalmic 10 µg generation 1 administered in the study eye on Day 1. One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
  Interventions: Drug: bimatoprost 10 µg generation 1; Drug: bimatoprost 0.03%

INTERVENTIONS:
Drug: bimatoprost 20 µg generation 2 — Single dose of bimatoprost ophthalmic administered in the study eye on Day 1.
  Arms: bimatoprost 20 µg generation 2, bimatoprost 0.03%
Drug: bimatoprost 15 µg generation 2 — Single dose of bimatoprost ophthalmic administered in the study eye on Day 1, and once between 90 days and 12 months after the first dose (if applicable).
  Arms: bimatoprost 15 µg generation 2, bimatoprost 0.03%
Drug: bimatoprost 10 µg generation 2 — Single dose of bimatoprost ophthalmic 10 µg generation 2 administered in the study eye on Day 1, and once between 90 days and 12 months after the first dose (if applicable).
  Arms: bimatoprost 10 µg generation 2, bimatoprost 0.03%
Drug: bimatoprost 6 µg generation 2 — Single dose of bimatoprost ophthalmic 6 µg generation 2 administered in the study eye on Day 1, and once between 90 days and 12 months after the first dose (if applicable).
  Arms: bimatoprost 6 µg generation 2, bimatoprost 0.03%
Drug: bimatoprost 15 µg generation 1 — Single dose of bimatoprost ophthalmic 15 µg generation 1 administered in the study eye on Day 1.
  Arms: bimatoprost 15 µg generation 1, bimatoprost 0.03%
Drug: bimatoprost 10 µg generation 1 — Single dose of bimatoprost ophthalmic 10 µg generation 1 administered in the study eye on Day 1.
  Arms: bimatoprost 10 µg generation 1, bimatoprost 0.03%
Drug: bimatoprost 0.03% — One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
  Other Names: LUMIGAN®

SUMMARY:
This study will evaluate the safety and efficacy of new ophthalmic formulations of bimatoprost in patients with open angle glaucoma and ocular hypertension. At least 3 dose strengths will be evaluated based on internal data review of each cohort. The study was planned to be conducted in 2 stages. Stage 1 was an open-label and Stage 2 was planned to be masked; however only Stage 1 was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma or ocular hypertension

Exclusion Criteria:

* Uncontrolled medical conditions
* Anticipated wearing of contact lenses during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-09-23 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (57):
- United States (36):
  - Sall Research Medical Center, Artesia, California
  - Shiley Eye Center, Hamilton Glaucoma Center, University of California, San Diego, La Jolla, California
  - Doheny Eye Institute, Los Angeles, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Shasta Eye Medical Group, Inc., Redding, California
  - Grutzmacher and Lewis, Inc., Sacramento, California
  - Pacific Eye Surgeons, San Luis Obispo, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Specialty Eye Care, Parker, Colorado
  - The Eye Associates of Manatee, Bradenton, Florida
  - Emory University, The Emory Eye Center, Atlanta, Georgia
  - Coastal Research Associates, Roswell, Georgia
  - Springfield Clinic, Springfield, Illinois
  - Glaucoma Consultants, Baltimore, Maryland
  - Tufts Medical Center/New England Eye Center, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Clinical Eye Research of Boston/ Charles River Eye Associates, Winchester, Massachusetts
  - Moyes Eye Center, Kansas City, Missouri
  - Northern New Jersey Eye Institute PA, South Orange, New Jersey
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Glaucoma Associates of NY, New York, New York
  - Rochester Ophthalmological Group PC, Rochester, New York
  - Charlotte Eye Ear Nose & Throat Associates, PA, Charlotte, North Carolina
  - Cornerstone Eye Care, High Point, North Carolina
  - James D. Branch, MD, Winston-Salem, North Carolina
  - Legacy Good Samaritan - Devers Eye Institute, Portland, Oregon
  - Scott & Christie and Associates, Cranberry Township, Pennsylvania
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - Keystone Research LTD, Austin, Texas
  - Glaucoma Associates of TX, Dallas, Texas
  - R and R Eye Research, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Focus Clinical Research, Salt Lake City, Utah
  - Spokane Eye Clinical Research, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
- Australia (2):
  - Melbourne Eye Specialists, Fitzroy
  - Eye Associates, Sydney New South Wales
- UZ Leuven, Campus St. Rafael, Dienst Oogheelkunde, Belgium
- Universidade Federal de São Paulo/Escola Paulista de Medicina/Hospital São Paulo Departamento de Oftalmologia, São Paulo, Brazil
- Canada (7):
  - A.C. S. Crichton Prof. Corp, Calgary, Alberta
  - Eye Care Center, Halifax, Nova Scotia
  - Anjema Eye Institute, Chatham, Ontario
  - Galen Eye Centre, Kingston, Ontario
  - Ivey Eye Institute, London, Ontario
  - Institut de l'œil des Laurentides, Boisbriand, Quebec
  - Clarity Eye Institute, Vaughan
- Staedtisches Klinikum Department of Opthalmology, Karlsruhe, Germany
- Israel (3):
  - Kaplan Medical Center, Rohovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Sam Rothberg Glaucoma Center,, Tel Litwinsky
- Philippines (3):
  - Asian Eye Institute, Makati City
  - Pacific Eye and Laser Institute (PELI), Makati City
  - St. Lukes Medical Center-Quezon City, Metro Manila
- Singapore National Eye Center, Singapore, Singapore
- Spain (2):
  - Valles Oftalmologia Recerca, Hospital General de Catalunya,, Sant Cugat del Vallès
  - Fundacion Oftalmologica Del Mediterraneo, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craven ER, Walters T, Christie WC, Day DG, Lewis RA, Goodkin ML, Chen M, Wangsadipura V, Robinson MR, Bejanian M; Bimatoprost SR Study Group. 24-Month Phase I/II Clinical Trial of Bimatoprost Sustained-Release Implant (Bimatoprost SR) in Glaucoma Patients. Drugs. 2020 Feb;80(2):167-179. doi: 10.1007/s40265-019-01248-0. PMID 31884564
- [Derived] Medeiros FA, Sheybani A, Shah MM, Rivas M, Bai Z, Werts E, Ahmed IIK, Craven ER. Single Administration of Intracameral Bimatoprost Implant 10 microg in Patients with Open-Angle Glaucoma or Ocular Hypertension. Ophthalmol Ther. 2022 Aug;11(4):1517-1537. doi: 10.1007/s40123-022-00527-6. Epub 2022 May 28. PMID 35643967

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 1, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 1, Bimatoprost 0.03%
Started | 15 | 21 | 21 | 18 | 11 | 23
Completed | 13 | 17 | 17 | 16 | 9 | 22
Not Completed | 2 | 4 | 4 | 2 | 2 | 1
Not completed — Other Reasons | 1 | 1 | 2 | 1 | 0 | 0
Not completed — Personal Reasons | 0 | 2 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 1, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 1, Bimatoprost 0.03% | Total
Number analyzed (Participants) | 15 | 21 | 21 | 18 | 11 | 23 | 109
Age, Customized [Number; unit: Participants]
  <45 years | 1 | 2 | 0 | 2 | 0 | 1 | 6
  45-65 years | 6 | 9 | 12 | 9 | 3 | 10 | 49
  >65 years | 8 | 10 | 9 | 7 | 8 | 12 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 9 | 12 | 5 | 13 | 56
  Male | 8 | 11 | 12 | 6 | 6 | 10 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Time-Matched Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: Baseline, Month 24
Population: Modified Intent-to-Treat: all treated patients with at least 1 IOP measurement at baseline and at least 1 postbaseline IOP measurement through Week 16. Excluding IOP assessments after rescue or retreatment.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Groups:
- Bimatoprost 15 μg Generation 1, Bimatoprost 0.03%: Single dose of bimatoprost ophthalmic 15 μg generation 1 administered in the study eye on Day 1. One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
- Bimatoprost 10 μg Generation 1, Bimatoprost 0.03%: Single dose of bimatoprost ophthalmic 10 μg generation 1 administered in the study eye on Day 1. One drop bimatoprost ophthalmic solution 0.03% (LUMIGAN®) administered in the non-study eye once daily every evening for up to 24 months.
Arm/Group | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 μg Generation 1, Bimatoprost 0.03% | Bimatoprost 10 μg Generation 1, Bimatoprost 0.03%
Number analyzed (Participants) | 15 | 21 | 21 | 18 | 11 | 23
Millimeters of Mercury (mmHg)
  Baseline Hour 0, | 26.57 (4.144) | 25.14 (2.967) | 24.48 (2.112) | 25.14 (3.609) | 23.73 (1.664) | 24.22 (2.104)
  Week 4, Hour 0: number analyzed (Participants) | 15 | 20 | 19 | 16 | 11 | 21
  Week 4, Hour 0 | -8.83 (3.750) | -7.80 (2.613) | -7.18 (3.250) | -7.09 (2.697) | -5.50 (3.507) | -7.33 (3.006)
  Week 12, Hour 0: number analyzed (Participants) | 12 | 21 | 18 | 17 | 11 | 22
  Week 12, Hour 0 | -7.92 (2.557) | -7.02 (3.215) | -6.82 (3.024) | -6.53 (4.091) | -5.95 (3.546) | -7.00 (2.899)
  Month 6, Hour 0: number analyzed (Participants) | 10 | 15 | 13 | 13 | 8 | 20
  Month 6, Hour 0 | -5.65 (3.652) | -6.50 (2.646) | -5.38 (3.015) | -6.81 (2.529) | -3.94 (4.170) | -5.40 (3.106)
  Month 12, Hour 0: number analyzed (Participants) | 6 | 7 | 6 | 8 | 5 | 7
  Month 12, Hour 0 | -9.00 (2.387) | -5.64 (2.824) | -6.00 (2.881) | -5.38 (3.091) | -5.80 (4.251) | -5.71 (2.138)
  Month 18, Hour 0: number analyzed (Participants) | 5 | 6 | 5 | 7 | 2 | 2
  Month 18, Hour 0 | -6.00 (3.464) | -6.92 (2.558) | -7.70 (3.493) | -6.93 (2.335) | -4.25 (0.354) | -9.75 (3.182)
  Month 24, Hour 0: number analyzed (Participants) | 4 | 5 | 5 | 5 | 1 | 1
  Month 24, Hour 0 | -5.75 (4.330) | -7.30 (2.019) | -7.40 (1.557) | -5.70 (2.197) | -8.50 (NA) — Standard Deviation is not applicable since there is only 1 patient. | -5.50 (NA) — Standard Deviation is not applicable since there is only 1 patient.

2. Secondary Outcome: Time-Matched Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measurement of the fluid pressure inside the study eye.
Time Frame: Baseline to Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 μg Generation 1, Bimatoprost 0.03% | Bimatoprost 10 μg Generation 1, Bimatoprost 0.03%
Number analyzed (Participants) | 15 | 21 | 21 | 18 | 11 | 23
Millimeters of Mercury (mmHg)
  Baseline, Hour 0 | 26.57 (4.144) | 25.14 (2.967) | 24.48 (2.112) | 25.14 (3.609) | 23.73 (1.664) | 24.22 (2.104)
  Week 4, Hour 0: number analyzed (Participants) | 15 | 20 | 19 | 16 | 11 | 21
  Week 4, Hour 0 | 17.73 (3.982) | 17.45 (2.032) | 17.55 (3.166) | 17.53 (2.661) | 18.23 (4.315) | 17.00 (2.748)
  Week 12, Hour 0: number analyzed (Participants) | 12 | 21 | 19 | 17 | 11 | 22
  Week 12, Hour 0 | 17.71 (2.996) | 18.12 (3.626) | 17.61 (2.289) | 18.03 (3.659) | 17.77 (2.970) | 17.23 (2.443)
  Month 6, Hour 0: number analyzed (Participants) | 10 | 15 | 13 | 13 | 8 | 20
  Month 6, Hour 0 | 19.10 (3.843) | 17.90 (3.785) | 19.35 (2.536) | 17.35 (2.135) | 19.44 (3.610) | 18.80 (3.282)

3. Secondary Outcome: Mean Diurnal IOP in the Study Eye
Description: IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0, 2, 4, 6, and 8 and averaged to determine the mean diurnal IOP.
Time Frame: Baseline, Month 6
Population: Modified Intent-to-Treat: all treated patients with at least 1 IOP measurement at baseline and at least 1 postbaseline IOP measurement through Week 16. Including IOP assessments after rescue or retreatment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 μg Generation 1, Bimatoprost 0.03% | Bimatoprost 10 μg Generation 1, Bimatoprost 0.03%
Number analyzed (Participants) | 15 | 21 | 21 | 18 | 11 | 23
mmHg
  Baseline | 23.38 (3.967) | 23.74 (3.411) | 23.02 (2.011) | 23.54 (5.121) | 20.84 (2.123) | 22.09 (2.521)
  Week 4: number analyzed (Participants) | 15 | 20 | 19 | 17 | 10 | 20
  Week 4 | 17.10 (4.584) | 16.59 (1.884) | 16.40 (2.529) | 17.35 (5.810) | 17.89 (2.038) | 16.88 (3.782)
  Week 12: number analyzed (Participants) | 15 | 21 | 19 | 17 | 11 | 23
  Week 12 | 17.34 (3.608) | 18.22 (3.294) | 17.33 (2.274) | 17.29 (3.199) | 17.12 (2.211) | 17.06 (2.604)
  Month 6: number analyzed (Participants) | 14 | 20 | 19 | 17 | 10 | 23
  Month 6 | 19.79 (4.498) | 18.51 (3.539) | 18.94 (2.879) | 16.71 (1.879) | 18.13 (3.080) | 18.55 (3.632)

4. Secondary Outcome: Time to Rescue Treatment or Re-Treatment in the Study Eye
Description: Time to rescue treatment or the second treatment in the generation 2 groups is defined as the time between the first treatment and the second treatment in the study eye.
Time Frame: 24 Months
Population: Modified Intent-to-Treat: all treated patients with at least 1 IOP measurement at baseline and at least 1 postbaseline IOP measurement through Week 16
Measure: Median (Full Range); unit: Days
Arm/Group | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 μg Generation 1, Bimatoprost 0.03% | Bimatoprost 10 μg Generation 1, Bimatoprost 0.03%
Number analyzed (Participants) | 15 | 21 | 21 | 18 | 11 | 23
Days | 328 [44 to 400] | 265 [119 to 534] | 273 [98 to 351] | 391.5 [13 to 553] | 411 [139 to 555] | 237 [2 to 611]

ADVERSE EVENTS:
Description: The Safety Population included all patients who received treatment and was used to assess adverse events and serious adverse events.
Arm/Group | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% | Bimatoprost 15 µg Generation 1, Bimatoprost 0.03% | Bimatoprost 10 µg Generation 1, Bimatoprost 0.03%
Serious Adverse Events (participants affected / at risk) | 0/15 | 3/21 | 6/21 | 4/18 | 3/11 | 3/23
Other Adverse Events (participants affected / at risk) | 12/15 | 16/21 | 17/21 | 15/18 | 8/11 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% (N=15) | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% (N=21) | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% (N=21) | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% (N=18) | Bimatoprost 15 µg Generation 1, Bimatoprost 0.03% (N=11) | Bimatoprost 10 µg Generation 1, Bimatoprost 0.03% (N=23)
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Allergy to Arthropod Sting (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Mantle Cell Lymphoma Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 20 µg Generation 2, Bimatoprost 0.03% (N=15) | Bimatoprost 15 µg Generation 2, Bimatoprost 0.03% (N=21) | Bimatoprost 10 µg Generation 2, Bimatoprost 0.03% (N=21) | Bimatoprost 6 µg Generation 2, Bimatoprost 0.03% (N=18) | Bimatoprost 15 µg Generation 1, Bimatoprost 0.03% (N=11) | Bimatoprost 10 µg Generation 1, Bimatoprost 0.03% (N=23)
Conjunctival Hyperaemia (Eye disorders) | 7 | 8 | 7 | 8 | 1 | 7
Foreign Body Sensation in Eyes (Eye disorders) | 4 | 2 | 3 | 4 | 2 | 3
Dry Eye (Eye disorders) | 3 | 1 | 1 | 0 | 1 | 2
Eye Pain (Eye disorders) | 3 | 4 | 4 | 1 | 2 | 3
Punctate Keratitis (Eye disorders) | 3 | 2 | 3 | 2 | 1 | 1
Conjunctival Haemorrhage (Eye disorders) | 2 | 4 | 3 | 3 | 1 | 5
Growth of Eyelashes (Eye disorders) | 2 | 1 | 1 | 1 | 0 | 0
Iris Hyperpigmentation (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 2 | 3 | 4 | 0 | 2 | 3
Vision Blurred (Eye disorders) | 2 | 2 | 2 | 2 | 1 | 3
Anterior Chamber Flare (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 1 | 1 | 1 | 0
Conjunctival Oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 1
Corneal Disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema of Eyelid (Eye disorders) | 1 | 1 | 1 | 1 | 0 | 2
Eyelid Margin Crusting (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eyelid Oedema (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 2
Eyelid Pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Eyelid Retraction (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eyelid Pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 1 | 5 | 3 | 1 | 1 | 4
Macular Cyst (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ocular Discomfort (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Optic Disc Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retinal Vein Occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 1 | 1 | 2 | 2 | 1
Anterior Chamber Inflammation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Corneal Opacity (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 2
Eye Pruritus (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 4
Iris Adhesions (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lid Margin Discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Orbit Atrophy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Corneal Oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hyphaema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Iritis (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 2
Lagophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Posterior Capsule Opacification (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Eyelid Ptosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 3
Vitreous Detachment (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 2
Intraocular Pressure Increased (Investigations) | 4 | 2 | 2 | 1 | 2 | 2
Blood Cholesterol Increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Gamma-glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood Potassium Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Heart Rate Irregular (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood Urine Present (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 3 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Progressive Multifocal Leukoencephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 1
Visual Field Defect (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Allergic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 2
Allergy to Arthropod Sting (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 0
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Transfusion Related Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Aqueous Humour Leakage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Corneal Dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mantle Cell Lymphoma Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.